CLINICAL TRIAL: NCT06815718
Title: Observational Study Evaluating the viQtor for Early Detection of Clinical Deterioration in Post-ICU Patients on General Wards
Acronym: ViQtor
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Michael Cornelis van Herwerden, Principal Investigator, Erasmus Medical Center
Other Study IDs: MEC-2024-0647
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Early Warning Score; Monitoring; Telemedicine-Based Education; Readmission; Rapid Response System
Keywords: Early Warning; EWS; Telemonitoring; continuous monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Telemonitoring group: Group wearing the ViQtor telemedicine solution for continuous monitoring

SUMMARY:
Rationale Following ICU discharge, intermittent vital sign monitoring may delay timely recognition of clinical deterioration and lead to unnecessary readmissions. This study proposes the use of the viQtor continuous monitoring device to measure pulse rate (PR), respiratory rate (RR), oxygen saturation (SpO2) and the activity index in post-ICU patients on general wards. The primary aim is to develop a continuous Early Warning Score (c-EWS), determine its optimal cut-off values. The secondairy outcome will be a comparison with the Modified Early Warning Score (MEWS). In addition, patient and nurse satisfaction, as well as technical feasibility, will be assessed.

DETAILED DESCRIPTION:
Objective(s) Primary: To develop and optimize a c-EWS using viQtor data for early detection of clinical deterioration in post-ICU patients.

Secondary: To evaluate the c-EWS's predictive accuracy relative to MEWS, to assess user satisfaction (patients and nurses), and to determine the technical feasibility of the viQtor device.

Study type This is a single-center prospective observational cohort study at general wards in post-discharge ICU patients.

Study population A single-center prospective observational cohort study will include approximately 180 post-ICU patients and 20 nurses at the Erasmus MC.

Methods Over a four-month period (winter/spring 2024-2025), patients transferred from the ICU to a general ward will wear the viQtor device for up to 5 days. Concurrent standard care involves MEWS measurements three times daily. No clinical decisions will be based on viQtor measurements, ensuring no interference with standard care. The c-EWS will be retrospectively derived and assessed using ROC analyses to determine optimal cut-off values. Comparisons with MEWS will be descriptive. Patient feedback will be collected via a brief questionnaire at discharge, and a semi-structured focus group with participating nurses will provide insights into user experiences.

Burden and risks The wearable viQtor device is noninvasive, comfortable, and worn continuously without affecting patient care or activities. Minor skin irritation is the only anticipated risk. Nurses' participation is limited to the focus group.

Recruitment and consent Patients will be screened in the last 48 hours of their ICU stay. Following informed consent, the viQtor device will be applied at the moment of transfer to the general ward. All participants will be fully informed about study procedures, potential risks, and their right to withdraw. Nurses will be invited via email to participate in the focus group and will provide informed consent before participation.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Written informed consent is obtained from the patient
* Expected hospitalization time after ICU discharge of 2 days or longer

Exclusion Criteria:

* The patient is unable to communicate in Dutch or English
* The patient has an allergy to metal or plastics (as the viQtor device contains these materials)
* The patient has significant deformities, swelling, irritation, degenerative changes, local infection, ulceration, skin lesions, or edema of the upper arms.
* The patient has tattoos on both upper arms where the device's PPG sensor would be placed
* The patient experiences tremors/and or convulsions affecting the upper arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted at Erasmus MC and will include 180 hospitalized adults (aged 18 years and older) who have received ICU care and are subsequently transferred to a general ward within the Erasmus MC.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Development and Validation of a Continuous Early Warning Score (c-EWS) for Detecting Clinical Deterioration in Post-ICU Patients Using the viQtor System | From enrollment to the end of monitoring in 5 days
  A continuous early warning score (c-EWS) will be developed using the viQtor system to detect clinical deterioration in post-ICU patients on the general ward. Clinical deterioration is defined as an ICU consultation or a Rapid Response Team intervention. The optimal cut-off values for the c-EWS will be identified and evaluated using Receiver Operating Characteristic (ROC) curves and the Area Under the Curve (AUC) values.

SECONDARY OUTCOMES:
Predictive Accuracy of c-EWS vs. MEWS for ICU Consultation or Rapid Response Team Intervention | 5 days
  The predictive accuracy of the optimized continuous Early Warning Score (c-EWS) compared to the Modified Early Warning Score (MEWS) in predicting ICU consultation or Rapid Response Team (RRT) intervention will be assessed using descriptive statistics.
Predictive Accuracy of c-EWS vs. MEWS for In-Hospital Cardiac Arrest, ICU Readmission, and Hospital Mortality | From enrollment to the end of monitoring (maximum 5 days).
  The predictive accuracy of the optimized c-EWS compared to the MEWS in predicting in-hospital cardiac arrest, ICU readmission, and hospital mortality will be assessed using descriptive statistics.
Predictive Accuracy of c-EWS in Detecting Clinical Deterioration Within 8 Hours of an Event | From enrollment to the end of monitoring (maximum 5 days).
  The ability of the viQtor system's c-EWS to detect clinical deterioration within the eight hours preceding a documented deterioration event will be evaluated using descriptive statistics.
Patient Acceptability of the viQtor System: Likert Questionnaire Results | end of monitoring after 5 days.
  Patient acceptability of using the viQtor solution will be assessed using a 5-point Likert questionnaire Responses will be analyzed descriptively to determine levels of acceptability.
Nurse Perspectives on the viQtor System: Thematic Analysis of Focus Group Results | At the end of the inclusion period
  Nurses' perspectives on the usability and feasibility of the viQtor system will be evaluated through semi-structured focus groups. Results will be thematically analyzed to identify key themes regarding user experience and implementation challenges.

CONTACTS AND LOCATIONS:
Overall Officials: Gerrie Prins, MD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided